#### SCREENING CONSENT

Title of Study: Phase I study of CDK 4-6 inhibitor PD-0332991 (palbociclib; IBRANCE) in children with recurrent, progressive or refractory central nervous system tumors

"You" refers to 'you' or 'your child' throughout this document. If you are the guardian of a minor or of a person under legal disability who is being asked to participate in this screening study, you may give consent on his/her behalf.

#### **INTRODUCTION:**

You have been asked to participate in a screening procedure for a research study. In order to decide whether or not you should agree to take part in the screening study, you should know enough about its risks and benefits to make your decision. This process is known as informed consent.

The study doctor or staff will explain the screening study to you and answer your questions about this testing. Screening study only include people who choose to take part. Before making your decision, please read the information below carefully. Please ask questions about anything you do not understand.

Once you understand the study, its risks and benefits, you will be asked to sign the form if you wish to take part. You will be given a copy to keep.

### Why is this study being done?

The purpose of this study is to perform a test on a sample of your tumor which was removed at the time of your surgery and has been stored in a hospital laboratory. This screening procedure is a test to see if you might qualify to take part in a main research study using a study drug called PD-0332991 (IBRANCE). By signing this consent form, you are not agreeing to participate in the main research study, but only agreeing to have this test done.

In order to participate in the main research study, your study doctor must assess whether your tumor tissue has a specific protein called Rb1 protein. This Rb1 protein is a protein that suppresses tumor growth. In certain tumors, cancer cells inactivate Rb1 protein so that it can no longer act as a tumor suppressor. However, over 60 percent of brain tumors in children still have Rb1 protein present and we want to find out whether your tumor has Rb1 protein or not. PD-0332991 (IBRANCE) is a capsule that prevents the inactivation of Rb1, thereby suppressing tumor growth.

You are being asked to participate in this study because you have a type of brain tumor other than diffuse pontine glioma (DIPG), medulloblastoma, or Atypical Teratoid Rhabdoid Tumor (ATRT) which has grown or come back after the usual treatment. Up to 55 people will be screened throughout the United States.

# What is involved in this screening procedure?

If you agree to have this screening test done, the study team will collect your date of birth to confirm your age, your tumor diagnosis, your height and weight and availability of your tumor tissue that was collected during a previous surgery.

The screening procedure will also include sending a piece of tumor tissue that was collected during a surgery to a laboratory at University of California, San Francisco (UCSF). Investigators from UCSF will look for the presence of Rb1 protein in the tumor tissue. If Rb1 protein is present, the study doctor or study nurse will discuss the main research study with you and you will be able to ask questions. If you are interested in taking part in the research study, you will be scheduled to have the rest of the eligibility procedures performed. You must meet all other eligibility criteria before you will able to participate in the main research study.

### How long will I be in the study?

Since this is just a screening procedure, your involvement in this study will be minimal. The screening test will be done as soon as possible after you sign this consent. The results will be given to your doctor who will discuss them with you and talk about the next steps.

### Can I stop being in the study?

Yes, you can decide to stop at any time. Tell the study doctor if you are thinking about stopping or decide to stop.

### What are the possible risks, side effects, and discomforts of this screening study?

Since your tumor tissue has already been collected during the surgery, there are no risks involved with this screening test.

### What are the benefits of participating in this study?

There are no benefits from having this tissue testing done other than to show if you might be able to participate in the main research study.

#### What other choices do I have if I do not take part in this study?

If you decide not to take part in this study, you will not be able to take part in the main research study. You do have choices. For example:

• you may choose to take part in a different study, if one is available

### Is my participation in this screening procedure voluntary?

Yes. The choice to take part in this study or not is yours.

#### Who will know about my participation in this screening study?

Every effort will be made to keep your study record private. However, we cannot guarantee total privacy. All records related to your involvement in this screening study will be stored in locked research files at: (hospital name). Your identity in these records will be indicated by a unique number rather than by your name, and the information linking these case numbers with your identity will be kept separate from the screening records.

Your personal information may be given out if required by law. If information from this study is published or presented at scientific meetings, your name and other personal information will not be used. Organizations that may look at and/or copy your medical records for screening, quality assurance, and data analysis include:

- Your referring physician.
- The local Institutional Review Board
- The Pediatric Brain Tumor Consortium, which coordinates this study
- The National Cancer Institute (NCI) and other government agencies, like the Food and Drug Administration (FDA), involved in keeping screening safe for people
- Representatives from pharmaceutical collaborators, such as the Pfizer company that supplies PD-0332991(IBRANCE)
- University of California, San Francisco

A description of this clinical trial may be available on http://www.ClinicalTrials.gov. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

### What are the costs of taking part in this study?

All costs associated with this screening procedure will be covered by the study budget. Neither you nor your insurance provider will be charged.

### Will I be paid if I take part in this screening procedure?

Participation in this screening procedure is voluntary. No payment for participation will be given.

#### What happens if I am injured because I took part in this study?

There is no risk of injury involved because this screening test will use previously collected tumor sample material.

# What are my rights if I take part in this study?

Taking part in the screening procedure is your choice. You may choose either to take part or not to take part in the screening procedure. No matter what decision you make, there will be no penalty to you and you will not lose any regular benefits. Your medical care will not be affected if you do not participate in this screening procedure. You can still get medical care from our institution.

### Who can answer my questions about the study?

You can talk to the study doctor about any questions or concerns you have about this study. Contact the study doctor (insert name of study doctor[s]) at (insert telephone number).

For questions about your rights while in this study, call the <u>(insert name of center)</u> Institutional Review Board (a group of people who review the research to protect your rights) at <u>(insert telephone number).</u>

# Where can I get more information?

You may call the National Cancer Institute's Cancer Information Service at:

1-800-4-CANCER (1-800-422-6237)

You may also visit the NCI Web site at http://cancer.gov/

For NCI's clinical trials information, go to: http://cancer.gov/clinicaltrials/. For NCI's general information about cancer, go to http://cancer.gov/cancerinfo/

You will get a copy of this form. If you want more information about this study, ask your study doctor.

### Signature

The above information has been explained to me and all of my current questions have been answered.

I understand that I am encouraged to ask questions about any aspect of this screening study during the course of this study, and that such future questions will be answered by a qualified individual or by the investigator(s) listed on the first page of this consent document at the telephone number(s) given. I understand that I may always request that my questions, concerns or complaints be addressed by a listed investigator.

By signing this form, I agree to participate in this screening study. A copy of this consent form will be given to me.

| PATIENT NAME:(Print Name) | | _ |
|-----------------------------------------------------------------|------|---|
| Signature of Patient or Parent or Legal Guardian or Next of Kin | Date | |
| Signature of 2 <sup>nd</sup> Parent or Legal Guardian | Date | |
| Signature of Investigator or Designee | Date | |
| Signature of Witness | Date | |

### **Model Consent Form**

# **Study Title for Study Participants:**

Testing PD-0332991 (IBRANCE) to prevent the tumor growth in children with brain tumors

# Official Study title for Internet Search on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>

PBTC-042: Phase I study of CDK 4-6 inhibitor PD-0332991 (palbociclib; IBRANCE) in children with recurrent, progressive or refractory central nervous system tumors

This form describes your participation in a clinical trial. "You" refers to 'you' or 'your child' throughout this document. If the research subject is a minor child, you may give consent on his/her behalf. A clinical trial is a type of research study. Clinical trials include only people who choose to take part. This consent form gives you information about this study, to be discussed with members of your study team.

Please take time to make the decision about whether to take part. Please discuss this decision with your family and friends. If there are any questions, ask your study doctor or health care team for more explanation.

# What is the usual approach to my type of cancer?

You are being asked to take part in this research study because you have a brain tumor that has grown or come back or not responded to the usual treatment. People who are not in a study are usually treated with surgery, chemotherapy, radiation or other investigational agents. Sometimes, combinations of these are used and your study doctor can explain which may be best for you. These treatments can reduce symptoms and may stop the tumor from growing for several months or more.

### What are my other choices if I do not take part in this study?

If you decide not to take part in this study, you have other choices. Please talk to your doctor about these other options. For example:

- You may choose to have the usual approach described above
- You may choose to take part in a different research study, if one is available
- Or you may choose not to be treated for cancer but you may want to receive comfort care to relieve symptoms.

### Why is this study being done?

Tumor cells grow and divide rapidly and uncontrollably. In normal cells, specific proteins called cyclin dependent kinases (CDK4 and 6) tightly control the process of cell division. Another protein called Rb1 also regulates cell division and stops the cells from dividing. By stopping cell division, the Rb1 protein suppresses tumor formation in normal cells. But in cancer, CDK4 and 6 are out of control and drive the cell to divide and form cancer. Tumor cells can sometimes inactivate Rb1 to help them divide continuously.

In this study, we are testing a study drug called PD-0332991 (IBRANCE) that works by inhibiting the CDK4 and 6 proteins. In animal studies, researchers have found that this drug works only if tumor cells have an intact Rb1 protein. Over 60 percent of brain tumors in children are likely to have an intact Rb1 protein. You have been approached for this study because your tumor has been identified to have an intact Rb1 protein. This drug is not FDA approved to treat brain tumors and is considered experimental.

PD-0332991 (IBRANCE) has been previously tested in adults only. This study is the first time this drug is being given to children. Therefore we are testing different doses of the drug to determine the maximum dose that can be safely given to children with cancer. Our hope is that PD-0332991 (IBRANCE) will be a more effective treatment for many types of childhood brain tumors. Approximately 42 - 50 people are expected to take part in this study throughout the United States. About 55 people will be screened in order to achieve this goal.

The purposes of this study are:

- 1. To find the highest dose of PD-0332991 (IBRANCE) that can be given without causing severe side effects in two study groups.
- 2. To learn what side effects may occur when PD-0332991 (IBRANCE) is given.
- 3. To learn how the body handles PD-0332991 (IBRANCE) by studying the levels of the drug in the blood.

# What are the study groups?

Patients will be divided into two groups based on the type and intensity of prior treatment received. To find the highest and safest dose, all study participants in each group will get different doses of the study drug PD-0332991 (IBRANCE). The first several study participants in each group will receive the lowest dose. If the initial dose level does not cause serious side effects, it will be given to other study participants at a higher dose. The doses will be increased for every group of study participants until side effects occur that require the dose to be lowered. If that dose level is safe, additional study participants will be included to receive PD-0332991 (IBRANCE) at the same dose level.

All study participants will get the study drug PD-0332991 (IBRANCE), in the form of oral capsules that should be taken with food. You will need to take PD-0332991 (IBRANCE) once a day for 21 days followed by 7 days break. This 4-week period is considered a course. You are encouraged to take your dose at the same time each day. It is important that you swallow the whole capsule (do not chew or crush). You should take plenty of water or take fluids to avoid dehydration if diarrhea occurs.

You will be given a medication diary to record the number of capsules you take each day and the time they are taken. You will also be asked to return any unused capsules and the bottles of PD-0332991 (IBRANCE) to your study doctor in each clinic appointment. If you vomit a dose of PD-0332991 (IBRANCE), you can re-dose if the capsule is seen intact in the vomited material. You will also be given a drug information handout and wallet card as a resource for yourself, caregivers and other health care providers.

# How long will I be in this study?

You will receive PD-0332991 (IBRANCE) for 26 courses (about 2 years). If you have benefited from receiving PD-0332991 (IBRANCE), and the study doctor agrees, you may be able to continue taking PD-0332991 (IBRANCE) for all 26 courses. Benefit means your disease is at least clinically and radiographically stable and you have not had any significant side effects. Your study doctor will continue to watch you for side effects and follow your condition for 30 days after your last dose of PD-0332991 (IBRANCE).

### What extra tests and procedures will I have if I take part in this study?

Most of the exams, tests, and procedures you will have are part of routine medical care for this type of cancer. However, there are some extra exams, tests and/or procedures that will need to be completed if you take part in this study.

## • Screening for Rb1 protein

If you have any type of CNS tumors other than DIPG, medulloblastoma, or ATRT, you will be asked to participate in the screening portion of this study. A screening test for presence or absence of Rb1 will be performed at a laboratory at University of California (UCSF). Your study doctor will send glass slides containing tumor tissue that was collected from a previous surgery to the lab. The tumor tissue will be stained to identify the Rb1 protein. Based on this analysis, which will take about 14 days, we will learn whether or not you are eligible for the study.

# • Electrocardiogram (EKG)

An electrocardiogram is a simple, painless test that records the heart's electrical activity. To assess the activity of your heart, your study doctor will do an EKG before you start the treatment. An EKG will also be performed 3 hours after you take the study drug PD-0332991 (IBRANCE) on days 1, 8 and 15 of Course 1. An EKG will also be done at these time points: day 1 of Courses 2 and 3, every 12 weeks and again at the end of treatment.

### • Eye exam

An eye exam will be performed by an ophthalmologist to make sure that you do not have or are not developing cataracts. It will be performed before you start the treatment and every 3 months while on study.

#### • Pharmacokinetics (PK) blood (required)

You are required to take part in this study because determining how the body handles this drug is an important part of the study. Your study doctor would like to learn how much PD-0332991 (IBRANCE) stays in the blood for specific time points after the drug is taken. A total of about 2 tablespoons (32 milliliters) of blood will be collected during the study.

Blood samples will be collected from you to determine how much of the drug stays in the blood. Less than ½ teaspoon (about 2 mL) of blood will be collected each time from your arm or central line before you start treatment and 30 minutes, 1, 2, 4, 8, 10 (optional), 24 and 48 hours after your first dose of PD-0332991 (IBRANCE). You will be told **NOT** to take PD-0332991 (IBRANCE) on Day 2 to collect the blood samples at 24 and 48 hour. Then, the same amount of blood will also be collected on Day 21 of Course 1 before you take PD-0332991 (IBRANCE) and 1, 2, 4, 8, 10 (optional) and 24 hours after you take PD-0332991 (IBRANCE).

The risks are the same for any blood sample collected from your line. If you don't have a central line, the most common risks related to drawing blood from your arm are brief pain and possibly a bruise.

Your privacy is very important to the researchers and they will make every effort to protect it. Your samples are sent to the research doctor but no information identifying you (such as your name or medical record number) will be sent. Samples will be identified by a unique code only. Information that identifies you will not be given to anyone, unless required by law. If research results are published, your name and other personal information will not be used.

You will not be billed for this required special study (Pharmacokinetics).

• PK blood after stopping Dexamethasone (steroid treatment given to decrease swelling in your brain) (optional)

This test is optional. The study doctor would like to find out how much PD-0332991 (IBRANCE) stays in the blood after you stop taking dexamethasone. If you choose to take part and have received dexamethasone during the required PK studies, the study doctor will collect serial blood samples at least 2 weeks after stopping dexamethasone, and after 2 weeks of continuous treatment with PD-0332991 (IBRANCE). Less than ½ teaspoon (about 2 mL) of blood will be collected for each sample.

# • Pharmacogenetics (optional)

If you choose to take part, a blood sample will be collected from you to determine if there are changes of certain genes that control how PD-0332991 (IBRANCE) is metabolized in the body. This test will require about 1 teaspoon (5 mL) of blood to be collected from your central line or a vein in your arm before you start the treatment.

• Pre-trial tumor material for genomics (optional)

Genomic research is research that studies the genes and their functions. Your blood and tumor cells contain genes, which are made up of DNA and which serve as the "instruction book" for cellular function. If you choose to take part, your study doctor would like to send a small piece of tumor material that is available from a previous surgery. The researchers will look for biological markers to help them understand the tumor better and how it might respond to the study drug.

### What will happen if I take part in this research study?

A study plan below shows how often these tests and procedures will be done while you are on this research study.

# Study Plan

| Test /Procedure | Pre-<br>therapy | Course 1 | Course 2 - Course 26 | Completion/<br>Discontinuation<br>Of Treatment |
|---|---|---|---|---|
| PHYSICAL ASSESSMENTS | | | | |
| Medical history, physical exam, vital signs, performance status, neurological exam | X | Every week | Every month | X |
| Blood counts | X | Every week | Every week | X |
| Blood Chemistries | X | Every week | Every month | X |
| Blood pregnancy test (for females who might be able to have children) | X | Before each course | | |
| Spinal tap (if needed) | X | | | |
| EKG | X | Day 1, 8, 15 | Day 1 of Course 2, 3, 6, 9, 12, 15, 18, 21 and 24 | X |
| Eye exam | X | | Course 3, 6, 9, 12, 15, 18, 21 and 24 | |
| Brain scan | X | | Course 2, 4, 6 and<br>then every 12<br>weeks | X |
| Spine scan (if needed) | X | | Same as Brain MRI if needed | X |
| Take PD-0332991 (IBRANCE) once a day; record in the pill diary | | X | X | |
| Optional research tests | | | | |
| Screening Pre-trial tumor materials for Rb1 testing (required for patients with all types of CNS tumors except DIPG, medulloblastoma, ATRT) | X | | | |
| Pharmacogenetics (if consented) | X | | | |
| Pharmacokinetics blood (required) | X | Day 1, 2, 3, 21 and 22 | | |
| PK blood after discontinuation of dexamethasone (if consented) | | Any time after stopping dexamethasone | | |
| Pre-trial tumor materials for Genomics (if consented) | X | | | |
| Tumor Tissue and blood for Biorepository (if consented) | X | | | |

# What possible risks can I expect from taking part in this study?

If you choose to take part in this study, there is a risk that:

- You may lose time at work, school or home and spend more time in the hospital or doctor's office than usual
- You may be asked sensitive or private questions which you do not normally discuss

The PD-0332991 (IBRANCE) used in this study may affect how different parts of your body work such as your liver, kidneys, heart, and blood. Your study doctor will be testing your blood and will address any changes that may affect your health.

There is also a risk that you could have side effects from PD-0332991 (IBRANCE).

Here are important points about side effects:

- Your study doctors do not know who will or will not have side effects.
- Some side effects may go away soon, some may last a long time, or some may never go away.
- Some side effects may interfere with your ability to have children.
- Some side effects may be serious and may even result in death.

Here are important points about how to make side effects less of a problem:

- Tell your study doctor if you notice or feel anything different so they can see if you are having a side effect.
- Your study doctor may be able to treat some side effects.
- Your study doctor may adjust the study drugs to try to reduce side effects.

Let your study doctor know of any questions you have about possible side effects. You can ask your study doctor questions about side effects at any time. The tables below show the most common and the most serious side effects that researchers know about. There might be other side effects that researchers do not yet know about. If important new side effects are found, your study doctor will discuss these with you.

#### Side effects of PD-0332991 (palbociclib; IBRANCE)

#### **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving palbociclib (PD-0332991), more than 20 and up to 100 may have:

- Anemia which may require blood transfusion
- Nausea
- Tiredness
- Infection, especially when white blood cell count is low

### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving palbociclib (PD-0332991), from 4 to 20 may have:

- Blurred vision, watering eyes
- Dry eye, skin
- Constipation, diarrhea, vomiting
- Sores in the mouth which may cause difficulty swallowing
- Fever
- Bruising, bleeding
- Loss of appetite
- Changes in taste
- Headache
- Nose bleed
- Hair loss, rash

**Reproductive risks:** You should not get pregnant, breastfeed, or father a baby while in this study. The effects of PD-0332991 (IBRANCE) used in this study could be very damaging to an unborn baby.

Women of childbearing potential must have a negative pregnancy test prior to study entry. Women of childbearing potential must agree to use an effective method of birth control during the study and for 97 days after completion of treatment. Check with your study doctor about what types of birth control, or pregnancy prevention, to use while in this study.

In animal studies, male reproductive organ effects were seen when PD-0332991 (IBRANCE) was given to rats and dogs for at least 3 weeks. The effects include decay of seminiferous tubule structure (tubes in the testes where sperm is produced) and a decrease in semen fluid secretion (ability of semen to flow). These effects were reported minimal to severe depending on the dose given. These toxicities were seen at drug levels that are used in clinical research studies. However, reversal of these effects were seen either partially or completely, at least 4 weeks after PD-0332991(IBRANCE) is stopped. It is currently unknown what these findings mean for patients treated with palbociclib over time. If you are a male patient and want to have children at a later time, we recommend that you preserve your sperm prior to the study entry. Male patients must agree to use effective contraception during the study and for 97 days after completion of treatment.

Routine studies in rats revealed that some of the animals developed cataracts (clouding of the eye lens) after being given PD-0332991 (IBRANCE) for 6 months. It is currently unknown what these findings mean for patients treated with PD-0332991 (IBRANCE) over time. You will have an eye examination done by your eye doctor to make sure that you do not have or are not developing cataracts before being registered on this study and every 3 months while on treatment.

### What possible benefits can I expect from taking part in this study?

Taking part in this study may or may not make your health better. This study may help doctors learn more about how PD-0332991 (IBRANCE) affects your cancer. This information could help future cancer patients.

# Can I stop taking part in this study?

Yes. You can decide to stop at any time. If you decide to stop for any reason, it is important to let your study doctor know as soon as possible so you can stop safely. If you stop, you can decide whether or not to let your study doctor continue to provide medical information to the organization running the study.

Your study doctor will provide any new information or changes in the study that may affect your health or willingness to continue in the study.

The doctor may decide to take you out of the study:

- If the side effects are too harmful to you
- If you need a treatment not allowed on this study
- If your tumor returns or grows
- If you do not follow the study rules
- If new information becomes available
- If the study is stopped by the sponsor, IRB or FDA

# What are my rights if I take part in this study?

Taking part in this study is your choice. No matter what your decision is, and even if your decision changes, there will be no penalty. You will not lose medical care or any legal rights.

For questions about you rights while taking part in this study, call the <u>(institution name)</u> Institutional Review Board (a group of people who review the research to protect your rights) at <u>(institution telephone number)</u>.

### What are the costs of taking part in this study?

PD-0332991 (IBRANCE) will be supplied at no charge while taking part in this study. It is possible that PD-0332991 (IBRANCE) may not continue to be supplied while you are on the study. Although not likely, if this occurs, your study doctor will talk to you about other options.

You or your health plan/insurance company will need to pay for all of the other costs of treating your cancer while in this study, including the cost of tests, procedures, or medicines to manage any side effects, unless your study doctor tells you certain tests are supplied at no charge. Before making a decision about participating in this study, you should check with your health plan or insurance company to find out exactly what they will pay for.

You will not be paid for taking part in this study.

### What happens if I am injured because I took part in this study?

If you are injured or hurt as a result of taking part in this study and need medical treatment, please tell your study doctor. The study sponsor will not offer to pay for medical treatment for injury. Your insurance company may not be willing to pay for study-related injury. If you have no insurance, you would be responsible for any costs.

If you feel this injury was a result of medical error, you keep all your legal rights to receive payment for this even though you are in a study.

### Who will see my medical information?

Your privacy is very important to us and the researchers will make every effort to protect it. Your personal information may be given out if required by law. However, the researchers will do their best to make sure that any information that is released will not identify you. Some of your health information, and/or information about your specimen, from this study will be kept in a central database for research.

There are organizations that may look at and/or receive copies of your medical records for research, quality assurance, and data analysis. Some of these organizations are:

- The study sponsor and the representatives from the pharmaceutical collaborator (Pfizer) who manufactures PD-0332991 (IBRANCE)
- The local Institutional Review Board, IRB, is a group of people who review the research with the goal of protecting people who take part in the study.
- The Pediatric Brain Tumor Consortium, who coordinates this study
- Federal agencies such as the Food and Drug Administration (FDA), the Office of Human Research Protections (OHRP) and the National Cancer Institute (NCI) in the U.S., and similar ones if other countries are involved in the study.

Coded patient data and images from brain scans will be transmitted over the Internet to be analyzed by other PBTC researchers. The PBTC has procedures (data encryption) in place to make electronic transmission of research information as secure as possible. The data security involves coding the data in a way that only the authorized receiver can decode the data. The method used to transfer information is more secure than many methods used by financial institutions when conducting business over the Internet.

### Where can I get more information?

You may visit the NCI Web site at http://cancer.gov/ for more information about studies or general information about cancer. You may also call the NCI Cancer Information Service to get the same information at: 1-800-4-CANCER (1-800-422-6237).

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Website will not include information that can identify you. At most the Website will include a summary of the results. You can search this Website at anytime

# Who can answer my questions about this study?

You can talk to your study doctor about any questions or concerns related to this study. Contact your study doctor (*Physician's name*) at (*Physician's telephone number*).

You will get a copy of this form. If you want more information about this study, ask your study doctor.

#### **Additional Studies Section:**

This part of the consent form is about optional studies that you can choose to participate. You will not get health benefits from any of these studies. The researchers leading these optional studies hope the results will help other people with cancer in the future.

You will not be billed for these optional studies. You can still take part in the main study even if you say "no" to any or all of these optional studies. If you sign up for but cannot complete any of the studies for any reason, you can still take part in the main study.

### What are the possible risks?

- 1. The most common risks related to drawing blood from your arm are brief pain and possibly a bruise.
- 2. There is a risk that someone could get access to the personal information in your medical records or other information researchers have stored.
- 3. There is a risk that someone could trace the information in a central database back to you. Even without your name or other identifiers, your genetic information is unique. The researchers believe the chance that someone will identify you is very small, but the risk may change in the future as people come up with new ways of tracing information.
- 4. There can also be a risk in knowing genetic information. New health information about inherited traits that might affect you or blood relatives could be found during a study. The researchers believe the chance these things will happen is very small, but cannot promise that they will not occur. In general, we will not give you any individual results from the study of the samples you gave us. This is because it will probably be a long time before we will know how to interpret the information accurately. In the rare instance that one of the genes tested might turn out to be an important risk factor for a disease, and having that information could allow you to take steps to prevent, detect earlier, or better treat that disease, we will ask you whether you want to know those results. If so, we will contact you and your doctor to discuss more testing.
- 5. Some of your genetic and health information may be placed in central databases that may be public, along with information from many other people. The data resulting from the genetic research may be deposited into a public or controlled access database made available to other researchers. Information that could directly identify you will not be included. However, people may develop ways in the future that would allow someone to link your genetic or medical information in our databases back to you. For example, someone could compare information in our databases with information from you (or a blood relative) in another database and be able to identify you (or your blood relative). It also is possible that there could be violations to the security of the computer systems used to store the codes linking your genetic and medical information to you.

# How will information be kept private?

Your privacy is very important to the researchers and they will make every effort to protect it. Here are just a few of the steps they will take:

1. When your sample(s) is sent to the researchers, no information identifying you (such as your name) will be sent. Samples will be identified by a unique code only.

- 2. The list that links the unique code to your name will be kept separate from your sample and health information.
- 3. Information that identifies you will not be given to anyone, unless required by law.
- 4. If research results are published, your name and other personal information will not be used.

# What are the possible benefits?

You will not benefit from taking part. The researchers, using the samples from you and others, might make discoveries that could help people in the future.

# What if I change my mind?

If you decide you no longer want research samples to be used, you can contact your study doctor in writing, <u>(insert name of study doctor)</u> who will let the researchers know. Then, any sample that remains in the bank will no longer be used and related health information will no longer be collected. Samples or related information that have already been given to or used by researchers will not be returned. If data has been submitted to a data repository, please include in your letter a request to retrieve your data.

# What if I have more questions?

If you have questions about the use of your samples for research, contact the study doctor, [Physician's name] at [Physician's telephone number].

For each of the optional studies below, please circle your response and then initial and date on the line provided.

### 1. Optional Sample Collection for research studies and storage:

Researchers are trying to learn more about cancer. Much of this research is done using samples from your tissue, blood, urine, or other fluids. Through these studies, researchers hope to find new ways to prevent, detect, treat, or cure health problems. Some of these studies may be about genes. Genes carry information about features that are found in you and in people who are related to you. Researchers are interested in the way that genes affect how your body responds to treatment. If you do not have tissues collected during or after treatment, ask your doctor how you can donate tissue in the future.

### i. Optional Sample Collection for Repository:

If you choose to take part in the sample collection for the repository, tumor tissue from a previous surgery is needed and a blood sample is strongly encouraged to provide stored genetic material from your tumor and your healthy tissue. The researchers ask your permission to store and use your samples and related health information (for example, your response to cancer treatment, results of study tests and medicines you are given) for future medical research. The future research that may be done is unknown at this time but may include genomic studies. These samples will be stored at the PBTC Central Review and Biorepository (PBTC CRB) where similar samples from other subjects are stored until requested for analysis.

| Version Date: 28 June | 2018 | |
|---|---|---|
| • | tumor tissue specimen collected and I agree that this tumory be used for the test described above. | r tissue and |
| YES | NO | |
| <u> </u> | blood specimen collected and I agree that this blood sample ed for the test described above. | and related |
| YES | NO | |
| If you choose to take used for the analysis researchers ask your percentage example, your respons for medical research. The I agree to have my specific to take used for the analysis research as a specific to take used for the analysis research. The I agree to have my specific to take used for the analysis of the analysis researchers as a specific to take used for the analysis researchers are a specific to take used for the analysis researchers. The analysis researchers are a specific to take used for the analysis researchers are a specific to take used for the analysis researchers are a specific to take used for the analysis researchers are a specific to take used for the analysis researchers. The analysis researchers are a specific to take used for the analysis researchers are a specific to take used for the analysis researchers. The analysis researchers are a specific to take us | le storage for future research: part, tumor material collected as a part of this study but not will be stored in the repository for future unspecified re ermission to store and use your samples and related health info e to cancer treatment, results of study tests and medicines you he research that may be done is unknown at this time. etimen collected and I agree that my specimen sample(s) and re ed for the laboratory study (ies) described above. | search. The<br>rmation (for<br>u are given) |
| YES | NO | |
| 2. Optional Laborat | ory studies | |
| If you choose to take p<br>determine if changes<br>through your body. T<br>medical care. This test<br>central line or arm bet<br>collected from your li<br>drawing blood from your<br>I choose to have my | genetic Study: art in this study, a blood sample will be collected from you for in certain genes are related to how PD-0332991 (IBRAN ne results of this test will only be used for research and not to will require about 1 teaspoon (5 mL) of blood to be collected fore you start the treatment. The risks are the same for any blue. If you don't have a central line, the most common risk ur arm are brief pain and possibly a bruise. | ICE) moves<br>o guide your<br>d from your<br>lood sample<br>as related to |
| YES | NO | |

NCI Protocol #: PBTC-042

# ii. PK blood after stopping Dexamethasone:

If you choose to take part and have received dexamethasone during the required PK studies, the study doctor will collect serial blood samples at least 2 weeks after stopping dexamethasone, and after 2 weeks of continuous treatment with PD-0332991 (IBRANCE). These samples will be collected at a routine clinic visit before you start treatment, and at 1, 2, 4, 8, 10 (optional) and at 24 hours after the dose. Less than ½ teaspoon (about 2 mL) of blood will be collected at each time point from your arm or central line. The risks are the same for any blood sample collected from your line. If you don't have a central line, the most common risks related to drawing blood from your arm are brief pain and possibly a bruise.

| from your urm are offer po | in and possiony a statist. | |
|---|---|---|
| · · | ecimen collected and I agree that my blood sample(s) and or the laboratory study described above. | d related |
| YES | NO | |
| iii. Pre-trial tumo | r material for genomics | |
| "instruction book" for the<br>doctor would like to sen<br>surgery. The researchers | mples contain genes, which are made up of DNA and servicells that make up our bodies. If you choose to take part, you a small piece of tumor material that is available from a will look for biological markers to help them understand the will not put you at risk as it will be taken from tumor already | our study<br>previous<br>e tumors |
| I agree that my tumor m described above. | aterial and related information may be used for the laborate | ory study |
| YES | NO | |
| If you chose to participate may choose to be contact samples. The results of to current study. | g incidental genetic findings in genetic testing of tumor samples as described in section 2 ted in the future if we find incidental genetic abnormalities nese studies or your choice will not affect your participation | s in your<br>on in the |
| I would like to be contact in my samples. | ed in the future if significant incidental genetic abnormalities a | are found |
| YES | NO | |

This is the end of the section about optional studies.

# **SIGNATURE**

| I have been given a copy of all pages of this form. I have a I understand the information and have had my questions answer main study and any additional studies where I circled 'yes'. | |
|---|---|
| PATIENT NAME:(Print Name) | |
| Signature of Patient or Parent or Legal Guardian or Next of Kin | Date |
| Signature of 2nd Parent or Legal Guardian | Date |
| Signature of Investigator or Designee | Date |
| Signature of Witness | <br>Date |